CLINICAL TRIAL: NCT00070694
Title: An Investigation of the Antidepressant Efficacy of the 5-HT2A Antagonist, M100907 in Combination With Escitalopram in Treatment Resistant Depression
Brief Title: An Investigation of the Antidepressant Efficacy of the 5-HT2A Antagonist, M100907, in Combination With Citalopram in Treatment Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030315; 03-M-0315
Record Dates: First submitted 2003-10-06; First posted 2003-10-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-10

CONDITIONS: Depressive Disorder
Keywords: Affective Disorders; Refractory; Augmentation; Polysomogram; Combination Therapy; Affective Disorder; Depression; Major Depression
MeSH Terms: conditions — Depressive Disorder; Mood Disorders; Depression; Depressive Disorder, Major

INTERVENTIONS:
Drug: MDL100.907

SUMMARY:
This study will examine whether a highly specific and powerful 5-hydroxytryptamine 2A (5-HT2A) antagonist, M100907, combined with escitalopram, is responsible for an antidepressant effect. Major affective disorders are common and can be chronic and life threatening. Yet as many as 50 to 75 percent of patients get only a partial response to the use of antidepressants. Some do not respond to medications in the category of serotonin reuptake inhibitors (SSRIs)-or they experience side effects that sharply interfere with daily life. This study will determine the extent to which M100907 improves sleep and improves fatigue in people who are treated, and how it reduces cognitive impairment, that is, limitations to awareness, in the depressive syndrome. It will also look at allele frequencies as being covariates in the analysis and to collect data.

Patients 18 to 65 years of age who meet the criteria for major depression, without psychotic features, may be eligible for this study. Women of childbearing potential must be using two medically accepted contraception methods and must agree to a (Beta)-HCG (human chorionic gonadotropin, a polypeptide hormone produced by the human placenta) test at the screening and at several intervals.

In random groups, participants will receive treatment with escitalopram and either M100907 or a placebo. The timing of escitalopram can be adjusted to manage side effects. If already taking any other medications for psychiatric purposes, participants will be tapered from those medications and monitored.

Participants will also undergo the following tests and procedures:

* Test of vital signs, lying and standing
* Physical exam
* 12-lead electrocardiogram (SCG)
* Psychiatric examination for screening
* Thyroid screening
* Collection of blood for chemistry and hematology
* Hepatitis B and C/HIV screening
* Beta-HCG pregnancy test, if applicable
* Urine drug screening
* Urinalysis
* Tests using the Hamilton Depression Rating Scale and the Montgomery-Asburg Depression Rating Scale
* Use of the Antidepressant Treatment History

A sleep study will be conducted during the steady state period and again toward the end of the double blind treatment period. Each study will involve 2 consecutive nights of polysomnographic recording done by an EEG technologist experienced in using the technique.

DETAILED DESCRIPTION:
Major Affective Disorders are common and often chronic life threatening illnesses. Furthermore a significant fraction of patients do not respond to treatment with serotonin reuptake inhibitors (SSRI's), have only a partial response with continued significant morbidity and functional impairment, or suffer from drug induced side effects that decrease the individuals' quality of life. Side effects from SSRI's include gastrointestinal symptoms, anxiety, sleep disturbance, and sexual dysfunction. Evidence from recent clinical trials and preclinical studies suggests that blockade of 5-HT2 receptors may have antidepressant effects when combined with reuptake blockade of serotonin at serotonin transporters. In order to better determine whether 5-HT2A receptors are responsible for this effect we propose to study the highly specific and potent 5-HT2A antagonist, M100907, in combination with escitalopram in SSRI resistant major depression.

Subjects aged 18-65 will be studied who prospectively are shown to be treatment resistant to the SSRI escitalopram. Subjects will be randomized in a double-blind fashion to receive continued open treatment with escitalopram+M100907 or continued escitalopram+placebo. Subjects will have weekly mood and safety ratings during this randomized period for four weeks. At that time subjects who were initially randomized to placebo (and are non-responders) will be switched to active drug for four weeks of randomized treatment while the active group continues an additional four weeks of combination therapy. Those meeting remission criteria will be eligible to extend therapy in open treatment with the combination therapy for an additional period of up to 6 months.

Due to the potential for M100907 to improve sleep architecture in general and slow wave sleep in particular, sleep will be studied using polysomnographic methods before and after randomization. Sleep disturbance is also a well-known side effect of SSRI's, and the addition of M100907 may improve sleep disturbance related to the affective disorder itself or to iatrogenic SSRI effects on sleep. Examination of improvement in sexual side effects, gastrointestinal side effects, headache frequency, and anxiety will also be investigated in the comparison of addition of M100907 versus placebo in escitalopram treated subjects. DNA samples will be collected for neurotransmitter-related genetic polymorphisms for covariance.

Finally, 5-HT2A receptors on cortical apical dendrites sit in a crucial location to influence cognitive processing and excitatory transmission. Since some 5-HT2A antagonists can lead to a down-regulation of 5-HT2A receptors and their altered distribution, as well as increased prefrontal cortical monoamine levels, neuropsychological testing to compare between and within subjects treated with M100907 and placebo may increase our understanding of the importance of serotonin receptors in cognition and depression. Subjects will be studied neuropsychologically before and twice following randomization. If M100907 enhances cognition in depression this would be an important advance given the high rates of impairment in functioning and residual cognitive difficulties observed in patients with depression.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects meeting all of the following criteria will be considered for enrollment into the study:

Men or women, 18 to 65 years of age.

A woman of childbearing potential must be using two medically accepted means of contraception. This can include an oral or other hormonal contraceptive started at least 4 weeks prior to randomization plus a barrier method such as condoms or two barrier methods combined. Surgical sterilization of the subject or their partner is also considered acceptable. Hormonal therapies should be in place at least 4 weeks prior to randomization (V8). Women of childbearing potential must agree to a beta test at screening and during Visits 5, 7, 8, 9, 11 and 13 through 16.

Each subject must have a level of understanding sufficient to agree to all tests and examinations required by the protocol.

Subjects must be considered reliable (i.e., based on clinical judgment of the investigator the subject is able and willing to cooperate with study procedures (including compliance with medication, use of birth control appropriately, and attend study visits, etc).

Each subject must understand the nature of the study and must sign an informed consent document.

Subjects must fulfill the criteria for major depression, without psychotic features as defined in DSM-IV based on clinical assessment and confirmed by structured diagnostic interview SCID-P.

Subjects must have an initial score at Visit 1 and Visit 2 of at least 20 on the HAM-D (17).

Subjects must have a total score of HAM-D at the end of the 6th week of escitalopram prospective screening of at least 17 (visit 5).

Current major depressive episode of at least 4 weeks duration and for the current episode of major depression has a history of failure to respond to at least 4 weeks of any antidepressant medication such as SSRI, Wellbutrin, nefazodone/trazadone, MAOI, or venlafaxine/duloxetine at an adequate or clinically customary dose for antidepressant purposes prior to entering escitalopram screening. Informed consent must be obtained in writing for all subjects at enrollment into the study.

EXCLUSION CRITERIA:

Subjects presenting with any of the following will not be included in the study:

No subjects who have previously been treated with the investigational product (M100907) will be enrolled in this study.

Participation in a clinical trial of another investigational (nonmarketed) drug within 1-month (30 days) prior to study Visit 1.

Female subjects who are either pregnant or breast-feeding or who do not appear reliable to use adequate contraception.

Clinically significant cardiovascular, hepatic, endocrinologic (including but not limited to diabetes and uncorrected hypothyroidism or hyperthyroidism), neurological (including but not limited to epilepsy, stroke and sleep apnea), or other major systemic disease making implementation of the protocol or interpretation of the study results difficult

Subjects with one or more past seizures without a clear and resolved etiology.

DSM-IV substance abuse (except nicotine and caffeine) within the past 90 days and substance dependence within the past 2 years.

Treatment with a reversible monoamine oxidase inhibitor, guanethidine, or guanadrel within 1 week prior to Visit 2.

Treatment with any other concomitant medication with primarily CNS activity, other than specified in Appendix 2 1 day prior to randomization.

Subjects are excluded if greater than four failed antidepressant trials in the past not including escitalopram (adequate dose and duration) during the index episode of major depression. An adequate trial is defined as 6 weeks of treatment with the antidepressant at a dosage considered therapeutic 159. The doses considered therapeutic are for fluoxetine 20-80 mg/day, paroxetine 20-60 mg/day, sertraline 100-200 mg/day, citalopram 20-40 mg/day, escitalopram 10-20 mg/day, fluvoxamine 100-300 mg/day, bupropion 300-450 mg/day, and venlafaxine 75-375 mg/day.

Failure to respond to drugs with a 5-HT2 mechanism when added to SSRI including nefazodone, trazodone, mirtazapine/mianserin, SSRI + atypical neuroleptics (clozapine, risperidone, olanzapine, ziprasidone) at therapeutic doses for 4 weeks or longer. (the SSRI must be at clinically appropriate doses and the 5-HT2 antagonist must be at doses that antagonize a significant % of receptors (trazadone greater than 125 mg, nefazodone greater than 300 mg, mirtazapine greater than 30 mg, clozapine greater than 50 mg, risperidone greater than .5 mg, olanzapine greater than 5mg, ziprasidone greater than 20 mg).

Treatment with electroconvulsive therapy (ECT) within 3 months prior to Visit 2.

Current diagnosis of schizophrenia or other psychotic or bipolar disorder as defined in the DSM-IV.

Judged clinically to be at serious risk of suicide based on HAM-D suicide item rating plus direct clinical questioning and assessment.

History of drug or alcohol dependence criteria in the last 2 years.

Hepatic enzyme elevation greater than 2X normal

Subjects who are taking drugs that could potentially interact with M100907 via the cyp 3A4 isoenzyme.

Subjects with a corrected Q-T ECG interval greater than 450 for males and 470 for females on screening ECG (Bazett correction)

History of hypersensitivity to the investigational products or to drugs with similar chemical structures.

Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol. Excluded meds: Treatment with CYP 3A4 inhibitors (macrolide antibiotics, itraconazole, indinivir, ritinivir, ketoconazol, verapamil, propoxyphene, fluoxetine) or inducers (rifampicin, carbamazepine, phenobarbitol, phenytoin). Treatment with sedative hypnotics or drugs with 5-HT2A or 5-HT3 activity (clozapine, risperidone, olanzapine, quetiapine, trazodone, nefazodone, mianserin, mirtazapine, cyproheptadine, ondansetron, granisetron, dolasetron). Treatment with drugs that are known to significantly prolong the QT interval of the ECG.

Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.

Subjects unlikely to comply with protocol, (e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study).

Subjects will not be allowed to receive psychotherapy during the trial..

Subjects may be included in the study only if they meet all of the inclusion and none of the exclusion criteria. The investigator and Aventis must approve any waiver of these inclusion and exclusion criteria on a case-by-case basis prior to enrolling the subject. Both Aventis and the investigator must document this. No subject will be allowed to enroll in this study more than once. The essential inclusion criteria for entry are subjects who have at least moderate level of major depression (HAM-D = 20) who do not have psychotic depression and are resistant to treatment based on both retrospective and prospective rating are treatment refractory to specified antidepressants. Subjects are excluded who have failed antidepressants of similar mechanism to M100907. Female subjects must use two forms of birth control and subjects will be excluded based on medical criteria outlined in the full list of inclusion and exclusion criteria.

No subjects who have previously been treated with the investigational product will be enrolled in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96
Dates: Start 2003-09; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Viguera AC, Baldessarini RJ, Friedberg J. Discontinuing antidepressant treatment in major depression. Harv Rev Psychiatry. 1998 Mar-Apr;5(6):293-306. doi: 10.3109/10673229809003578. PMID 9559348
- [Background] Solomon DA, Keller MB, Leon AC, Mueller TI, Shea MT, Warshaw M, Maser JD, Coryell W, Endicott J. Recovery from major depression. A 10-year prospective follow-up across multiple episodes. Arch Gen Psychiatry. 1997 Nov;54(11):1001-6. doi: 10.1001/archpsyc.1997.01830230033005. PMID 9366656
- [Background] Thase ME, Entsuah AR, Rudolph RL. Remission rates during treatment with venlafaxine or selective serotonin reuptake inhibitors. Br J Psychiatry. 2001 Mar;178:234-41. doi: 10.1192/bjp.178.3.234. PMID 11230034